CLINICAL TRIAL: NCT01321723
Title: A Double Blind, Randomized, Repeat Dose Parallel Group Study of Recombinant Human Parathyroid Hormone Analog Tablets, or Placebo Tablets, Compared to Open Label Forsteo® in Postmenopausal Women With Osteoporosis
Brief Title: Pharmacodynamics, Pharmacokinetics, Safety and Tolerability of PTH Analog Tablets in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unigene Laboratories Inc. (Industry)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UGL-OR1001
Record Dates: First submitted 2011-03-16; First posted 2011-03-23 (Estimated); Results first posted 2013-02-21 (Estimated); Last update posted 2013-03-01 (Estimated); Status verified 2013-01

CONDITIONS: Postmenopausal Osteoporosis
Keywords: Osteoporosis; Bone Diseases, Metabolic; Bone Diseases; Bone Density Conservation Agents
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis; Bone Diseases, Metabolic; Bone Diseases | interventions — parathyroid hormone (1-31); Teriparatide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- PTH analog tablet (Experimental): PTH(1-31) 5 mg tablet, once daily
  Interventions: Drug: PTH analog
- Placebo (Placebo Comparator): Placebo matching tablet, once daily
  Interventions: Drug: Placebo
- Forsteo (Active Comparator): Forsteo (teriparatide) 20 mcg SC Injection, once daily
  Interventions: Drug: Forsteo (Teriparatide)

INTERVENTIONS:
Drug: PTH analog — A recombinant 1-31 amino acid fragment of PTH.
  Other Names: PTH(1-31)
  Arms: PTH analog tablet
Drug: Placebo
  Arms: Placebo
Drug: Forsteo (Teriparatide) — A recombinant 1-34 amino acid fragment of PTH.
  Other Names: Forteo (US)
  Arms: Forsteo

SUMMARY:
This study is designed to provide information about the bone anabolic properties and absorption profile of Unigene's PTH Analog when administered as oral tablets over a period of 24 weeks to postmenopausal women with osteoporosis.

DETAILED DESCRIPTION:
The choice of a 24-week treatment period was based on published studies of PTH which demonstrate its potential to produce a statistically significant increase in BMD in patients with postmenopausal osteoporosis within that observation period.

ELIGIBILITY:
Inclusion Criteria:

* Healthy postmenopausal women (45-80 years old) with a diagnosis of osteoporosis

Exclusion Criteria:

* Use of estrogen or hormone replacement therapy
* Use of bisphosphonates, strontium ranelate or denosumab
* Use of parathyroid analogues or other bone metabolic agents
* Medical conditions which might alter bone metabolism
* Any known clinically significant disease affecting calcium metabolism or history of metabolic disorders including Paget's disease, osteogenesis imperfecta, or osteomalacia
* Impairment of thyroid function

Ages: 45 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christence S Teglbjaerg, MD, Principal Investigator — CCBR; Bettina S Nedergaard, MD, Principal Investigator — CCBR; Peter Alexandersen, MD, Principal Investigator — CCBR; Ivo Valter, MD, Principal Investigator — CCBR
Locations (4):
- Denmark (3):
  - CCBR, Aalborg
  - CCBR, Ballerup Municipality
  - CCBR, Vejle
- CCBR, Tallinn, Estonia

REFERENCES:
- [Result] Henriksen K, Andersen JR, Riis BJ, Mehta N, Tavakkol R, Alexandersen P, Byrjalsen I, Valter I, Nedergaard BS, Teglbjaerg CS, Stern W, Sturmer A, Mitta S, Nino AJ, Fitzpatrick LA, Christiansen C, Karsdal MA. Evaluation of the efficacy, safety and pharmacokinetic profile of oral recombinant human parathyroid hormone [rhPTH(1-31)NH(2)] in postmenopausal women with osteoporosis. Bone. 2013 Mar;53(1):160-6. doi: 10.1016/j.bone.2012.11.045. Epub 2012 Dec 9. PMID 23234813
- [Derived] Sturmer A, Mehta N, Giacchi J, Cagatay T, Tavakkol R, Mitta S, Fitzpatrick L, Wald J, Trang J, Stern W. Pharmacokinetics of oral recombinant human parathyroid hormone [rhPTH(1-31)NH(2)] in postmenopausal women with osteoporosis. Clin Pharmacokinet. 2013 Nov;52(11):995-1004. doi: 10.1007/s40262-013-0083-4. PMID 23719683

RESULTS

PARTICIPANT FLOW:
Groups:
- Forsteo (Teriparatide): Teriparatide : 20 mcg SC Injection, once daily.
- PTH Analog Tablets: PTH analog : 5 mg tablets, once daily.
- Placebo: Placebo : matching tablets, once daily
Period: Overall Study
Arm/Group | Forsteo (Teriparatide) | PTH Analog Tablets | Placebo
Started | 32 | 33 | 32
Completed | 27 | 28 | 28
Not Completed | 5 | 5 | 4
Not completed — Adverse Event | 3 | 5 | 2
Not completed — Withdrawal by Subject | 2 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Forsteo (Teriparatide) | PTH Analog Tablets | Placebo | Total
Number analyzed (Participants) | 32 | 33 | 32 | 97
Age Continuous [Mean (Standard Deviation); unit: years] | 66.5 (6.99) | 67.4 (3.95) | 66.1 (6.09) | 66.7 (5.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 33 | 32 | 97
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: % Change From Baseline BMD in L1-L4 Axial Lumbar Spine at Week 24
Time Frame: 24 weeks from baseline
Population: mITT Population: all subjects who received at least one dose of treatment and at least one post-baseline BMD value. Missing data imputation for patients who completed Week 12 but not the full 24-week period, data was imputed using the LOCF. No data imputation was performed for Week 24, if the Week 12 data was missing.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Forsteo (Teriparatide) | PTH Analog Tablets | Placebo
Number analyzed (Participants) | 30 | 28 | 27
percentage of change | 5.07 (3.543) | 2.21 (2.503) | -0.17 (2.739)

2. Post Hoc Outcome: Number of Participants With AEs as a Measure of Safety and Tolerability
Time Frame: 24 weeks
Population: Overall Summary of Adverse Events - Each subject with an event is counted only once although they may have several events.
Measure: Number; unit: participants
Arm/Group | Forsteo (Teriparatide) | PTH Analog Tablets | Placebo
Number analyzed (Participants) | 32 | 33 | 32
participants | 23 | 30 | 21

3. Secondary Outcome: % Change From Baseline in Bone Resorption Marker (CTx-1) at Week 24
Description: Serum collagen type I (CTx-1) fragments generated during osteoclastic bone turnover are biomarkers for bone resorption. β-CrossLaps electrochemiluminescent sandwich immunoassay was used.
Time Frame: 24 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Forsteo (Teriparatide) | PTH Analog Tablets | Placebo
Number analyzed (Participants) | 30 | 28 | 28
percentage of change | 113.32 (102.932) | 12.72 (36.547) | 15.13 (23.940)

4. Secondary Outcome: Systemic Absorption of PTH at Week 24
Description: AUC: (PTH analog tablets timepoints - baseline to 5.75 hours) (Forsteo injection timepoints - baseline to 2 hours)
Time Frame: 24 weeks
Measure: Mean (Standard Deviation); unit: pg* hr/mL
Arm/Group | Forsteo (Teriparatide) | PTH Analog Tablets
Number analyzed (Participants) | 27 | 28
pg* hr/mL | 152 (65.7) | 165 (180)

5. Secondary Outcome: % Change From Baseline in Bone Formation Marker (P1NP) at Week 24
Time Frame: 24 weeks from baseline
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Forsteo (Teriparatide) | PTH Analog Tablets | Placebo
Number analyzed (Participants) | 30 | 28 | 28
percentage of change | 210.07 (202.613) | 12.05 (37.055) | -1.75 (27.459)

ADVERSE EVENTS:
Time Frame: All AEs were recorded in the CRF during the course of the study. Serious adverse events (SAEs) were reported to the Sponsor within 24 hours of awareness.
Description: The occurrences of AEs were documented at each visit during the study.
Arm/Group | Forsteo (Teriparatide) | PTH Analog Tablets | Placebo
Serious Adverse Events (participants affected / at risk) | 1/32 | 2/33 | 2/32
Other Adverse Events (participants affected / at risk) | 23/32 | 30/33 | 21/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Forsteo (Teriparatide) (N=32) | PTH Analog Tablets (N=33) | Placebo (N=32)
Atrial flutter (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Forsteo (Teriparatide) (N=32) | PTH Analog Tablets (N=33) | Placebo (N=32)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 6 (6) | 2 (2)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 13 (13) | 6 (6)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 2 (2) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 3 (3) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Dizziness (Vascular disorders) | 3 (3) | 3 (3) | 2 (2)
Fatigue (General disorders) | 2 (2) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 3 (3) | 2 (2)
Hot flush (Vascular disorders) | 2 (2) | 1 (1) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 3 (3) | 0 (0)
Hypertension (Vascular disorders) | 1 (1) | 2 (2) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 4 (4) | 0 (0)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2)
Nasopharyngitis (Infections and infestations) | 3 (3) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 3 (3) | 5 (5) | 2 (2)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0) | 2 (2)
Presyncope (Cardiac disorders) | 0 (0) | 1 (1) | 2 (2)
Rhinitis (Infections and infestations) | 2 (2) | 1 (1) | 1 (1)
Syncope (Cardiac disorders) | 0 (0) | 4 (4) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No